CLINICAL TRIAL: NCT03316521
Title: Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of a Single Ascending Dose (SAD) and a Multiple Dose (MD) of the Complement Inhibitor AMY-101. A Prospective, Single-center, Open-label, First-In-Human (FIH) Clinical Study in Healthy Male Volunteers
Brief Title: First-In-Human Clinical Study of the C3 Complement Inhibitor AMY- 101 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amyndas Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMY-101/01
Record Dates: First submitted 2017-08-11; First posted 2017-10-20 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Complement Mediated Diseases
Keywords: complement inhibition; C3 complement inhibitor; AMY-101; Compstatin Cp40; Paroxysmal Nocturnal Hemoglobinuria (PNH); C3 glomerulopathy (C3G); Periodontal disease; Age-related macular degeneration (AMD); ABO incompatible kidney transplantation
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Periodontal Diseases; Macular Degeneration | interventions — AMY-101

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, open-label FIH study investigating the safety, tolerability, PK and PD after single and multiple doses of AMY-101 in healthy male volunteers. In the SAD part of the study, a single dose at ascending dose levels of AMY-101 will be administered to different cohorts, following a careful dose-escalation strategy. In the MD part of the study, multiple doses will be administered using different dosing intervals; the cohorts will include a minimum of four (4) subjects each. Additional subjects may be added in the cohorts if necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): In the SAD arm subjects will be sequentially included in one of up to six cohorts (dose levels). All cohorts will include at least four subjects each. Additional subjects may be added in any cohort if necessary.
  AMY-101 will be administered as a SQ or IV injection. Subjects in each cohort will be dosed sequentially, to allow for close safety monitoring. Between each cohort, safety data will be analyzed, evaluated and reviewed by the internal Safety Review Committee. Subsequent dose levels will be administered until either the maximum tolerated dose (MTD) or the study maximum dose (SMD) is reached based on specified dose escalation criteria.
  Interventions: Drug: AMY-101
- Multiple Dose (MD) (Experimental): Depending on the results of the SAD, multiple doses of AMY-101 will be administered at the dose which has been identified as the dose which saturates target C3, for a duration that results to an exposure level equivalent to the maximum exposure achieved in the SAD. The dose and dosing interval will be determined based on the PK data obtained in the SAD part of the study. Each MD cohort will include at least four subjects and may be expanded with additional subjects if necessary. Between each cohort, safety data will be analyzed, evaluated and reviewed by the internal Safety Review Committee.
  Interventions: Drug: AMY-101

INTERVENTIONS:
Drug: AMY-101 — AMY-101 is a selective inhibitor of complement activation, which binds to the complement component C3.

SUMMARY:
Safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a Single Ascending Dose (SAD) and a Multiple Dose (MD) of the complement inhibitor AMY-101. A prospective, single-center, open-label, First-In-Human (FIH) clinical study in healthy male volunteers.

DETAILED DESCRIPTION:
AMYNDAS is developing a novel peptidic complement inhibitor AMY-101, based on the third-generation compstatin analogue Cp40. AMY-101 is a selective inhibitor of complement activation in humans and in NHP. It binds to the complement component C3, the central "functional hub" that controls the upstream activation/amplification and downstream effector functions of complement. By binding to C3, AMY-101 inhibits the cleavage of native C3 to its active fragments C3a and C3b. As a consequence, the deposition of C3b, amplification via the alternative pathway and all downstream complement responses are prevented. AMY-101 is being developed to treat complement-mediated diseases, which are largely driven by aberrant C3 activation.

This first-in-human study of the C3-targeting complement inhibitor AMY-101 investigates the safety and PK/PD profile of AMY-101 in healthy male volunteers after Single Ascending Dose (SAD) and Multiple Doses (MD) using subcutaneous (SQ) or intravenous (IV) administration. The study is a prospective, single-center, open-label evaluation in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male subject aged 18-60 years, inclusive at the time of signing the informed consent.
3. Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 and weight at least 50 kg.
4. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Willing to use condom and contraceptive methods with a failure rate of < 1% to prevent pregnancy and drug exposure of a partner and to refrain from donating sperm from the date of dosing until three (3) months after dosing of the IMP.
6. Willing and able to complete all procedures according to the Protocol.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History of any Neisseria meningitidis infection
3. History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within the last 60 days prior to dosing.
4. History of latent or active tuberculosis, as assessed by the investigator based on chest X-ray and positive Quantiferon-TB Gold test.
5. History of complement deficiency.
6. History of any type of malignancy. However, completely resolved minor malignancies, at the discretion of the Investigator, may not be an exclusion criterion (for example: Non-Melanoma Skin Cancer).
7. Diagnosis of autoimmune, immunologic or rheumatologic disease (eg, systemic lupus erythematosus, rheumatoid arthritis).
8. Any clinically significant illness, medical/surgical procedure or trauma within four (4) weeks of the administration of IMP.
9. High CRP at screening (> 0.5 mg/dL).
10. Current evidence or history of bacterial, viral or fungal infection within 14 days prior to (first) dosing or longer according to the judgment of the investigator for e.g. viral infections including herpes simplex or herpes zoster.
11. Any current condition or risk, which, in the opinion of the Investigator, may interfere with the subject's participation in the study, poses an added risk for the subject, or confounds the assessment of the subject or outcome of the study
12. Any clinically significant abnormality in clinical chemistry, hematology, or urinalysis results at the time of screening, as judged by the Investigator.
13. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and/or Human Immunodeficiency Virus (HIV).
14. After 10 minutes supine rest abnormal vital signs defined as any of the following:

    * Systolic BP > 140 mm Hg
    * Diastolic BP > 95 mm Hg
    * HR < 40 or > 90 beats per minute
15. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormality in the resting ECG, as judged by the Investigator.
16. Any history of any allergy/hypersensitivity or anaphylactic reaction or on-going allergy/hypersensitivity. History of hypersensitivity to antibiotics or drugs with a similar chemical structure or class to AMY-101.
17. Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two (2) weeks prior to the administration of IMP, except the occasional intake of paracetamol/acetominophen (maximum 2000 mg/day; and not exceeding 3000 mg/week) or nasal decongestant without cortisone or antihistamine, at the discretion of the Investigator.
18. Administration of another new chemical entity (defined as a compound that has not been approved for marketing) or having participated in any other clinical study that included drug treatment within 30 day or 5 half lives of the last administration of the other IMP. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
19. Immunization with a live-attenuated vaccine one (1) month prior to the first administration of IMP.
20. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three (3) times per week is allowed before screening visit.
21. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
22. Positive screen for drugs of abuse at screening or on admission to the unit or positive screen for alcohol at screening or on admission to the unit prior to administration of the IMP.
23. Use of anabolic steroids.
24. Plasma donation within one (1) month of screening or any blood donation/blood loss > 450 mL during the three (3) months prior to screening.
25. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 21 days after treatment.

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUCt) after a single dose | Up to 14 days after treatment.
Area under the plasma concentration time curve from zero to infinity (AUC 0->∞) after a single dose | Up to 14 days after treatment.
Peak Plasma Concentration (Cmax) after single and multiple doses | Up to 14 days after treatment.
Time to Cmax (Tmax) after single and multiple doses | Up to 14 days after treatment.
Terminal elimination rate constant (lambdaz) after single and multiple doses | Up to 14 days after treatment.
Terminal half-life (T1/2) after single and multiple doses | Up to 14 days after treatment.
Total apparent clearance of drug from plasma/serum (CL/F) after single and multiple doses | Up to 14 days after treatment.
Volume of distribution (Vz) / fraction of drug absorbed (F) after single and multiple doses | Up to 14 days after treatment.
Area under the curve at steady state (AUCss) after multiple doses | Up to 14 days after treatment.
Activation of the classical complement pathway | Up to 14 days after treatment.
  CH50
Activation of the alternative complement pathway | Up to 14 days after treatment.
  AP50
Complement protein C3 plasma levels | Up to 14 days after treatment.
Complement protein C4 plasma levels | Up to 14 days after treatment.
Measurement of immune response (plasma protein electrophoresis - IgG,IgA, IgM) after single and multiple administrations of AMY-101. | Up to 14 days after treatment.
Investigation for anti-drug antibodies after single and multiple administrations of AMY-101. | Up to 14 days after treatment.
Measurement of lymphocyte subsets after multiple administrations of AMY-101. | Up to 14 days after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- HighPoint Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricklin D, Lambris JD. Complement in immune and inflammatory disorders: therapeutic interventions. J Immunol. 2013 Apr 15;190(8):3839-47. doi: 10.4049/jimmunol.1203200. PMID 23564578
- [Background] Ricklin D, Lambris JD. Complement in immune and inflammatory disorders: pathophysiological mechanisms. J Immunol. 2013 Apr 15;190(8):3831-8. doi: 10.4049/jimmunol.1203487. PMID 23564577
- [Background] Mastellos DC, Yancopoulou D, Kokkinos P, Huber-Lang M, Hajishengallis G, Biglarnia AR, Lupu F, Nilsson B, Risitano AM, Ricklin D, Lambris JD. Compstatin: a C3-targeted complement inhibitor reaching its prime for bedside intervention. Eur J Clin Invest. 2015 Apr;45(4):423-40. doi: 10.1111/eci.12419. Epub 2015 Mar 9. PMID 25678219
- [Background] Ricklin D, Lambris JD. Therapeutic control of complement activation at the level of the central component C3. Immunobiology. 2016 Jun;221(6):740-6. doi: 10.1016/j.imbio.2015.06.012. Epub 2015 Jun 10. PMID 26101137
- [Background] Reis ES, Mastellos DC, Yancopoulou D, Risitano AM, Ricklin D, Lambris JD. Applying complement therapeutics to rare diseases. Clin Immunol. 2015 Dec;161(2):225-40. doi: 10.1016/j.clim.2015.08.009. Epub 2015 Sep 1. PMID 26341313
- [Background] Mastellos DC, Ricklin D, Hajishengallis E, Hajishengallis G, Lambris JD. Complement therapeutics in inflammatory diseases: promising drug candidates for C3-targeted intervention. Mol Oral Microbiol. 2016 Feb;31(1):3-17. doi: 10.1111/omi.12129. Epub 2015 Oct 7. PMID 26332138
- [Background] Reis ES, DeAngelis RA, Chen H, Resuello RR, Ricklin D, Lambris JD. Therapeutic C3 inhibitor Cp40 abrogates complement activation induced by modern hemodialysis filters. Immunobiology. 2015 Apr;220(4):476-82. doi: 10.1016/j.imbio.2014.10.026. Epub 2014 Nov 3. PMID 25468722
- [Background] Mastellos DC, Ricklin D, Yancopoulou D, Risitano A, Lambris JD. Complement in paroxysmal nocturnal hemoglobinuria: exploiting our current knowledge to improve the treatment landscape. Expert Rev Hematol. 2014 Oct;7(5):583-98. doi: 10.1586/17474086.2014.953926. Epub 2014 Sep 2. PMID 25213458
- [Background] Risitano AM, Ricklin D, Huang Y, Reis ES, Chen H, Ricci P, Lin Z, Pascariello C, Raia M, Sica M, Del Vecchio L, Pane F, Lupu F, Notaro R, Resuello RR, DeAngelis RA, Lambris JD. Peptide inhibitors of C3 activation as a novel strategy of complement inhibition for the treatment of paroxysmal nocturnal hemoglobinuria. Blood. 2014 Mar 27;123(13):2094-101. doi: 10.1182/blood-2013-11-536573. Epub 2014 Feb 4. PMID 24497537
- [Background] Mastellos DC, Reis ES, Yancopoulou D, Hajishengallis G, Ricklin D, Lambris JD. From orphan drugs to adopted therapies: Advancing C3-targeted intervention to the clinical stage. Immunobiology. 2016 Oct;221(10):1046-57. doi: 10.1016/j.imbio.2016.06.013. Epub 2016 Jun 16. PMID 27353192
- [Background] Maekawa T, Briones RA, Resuello RR, Tuplano JV, Hajishengallis E, Kajikawa T, Koutsogiannaki S, Garcia CA, Ricklin D, Lambris JD, Hajishengallis G. Inhibition of pre-existing natural periodontitis in non-human primates by a locally administered peptide inhibitor of complement C3. J Clin Periodontol. 2016 Mar;43(3):238-49. doi: 10.1111/jcpe.12507. Epub 2016 Mar 3. PMID 26728318
- [Background] Hajishengallis G, Maekawa T, Abe T, Hajishengallis E, Lambris JD. Complement Involvement in Periodontitis: Molecular Mechanisms and Rational Therapeutic Approaches. Adv Exp Med Biol. 2015;865:57-74. doi: 10.1007/978-3-319-18603-0_4. PMID 26306443
- [Background] Hajishengallis G, Hajishengallis E, Kajikawa T, Wang B, Yancopoulou D, Ricklin D, Lambris JD. Complement inhibition in pre-clinical models of periodontitis and prospects for clinical application. Semin Immunol. 2016 Jun;28(3):285-91. doi: 10.1016/j.smim.2016.03.006. Epub 2016 Mar 24. PMID 27021500
- [Background] Zhang Y, Shao D, Ricklin D, Hilkin BM, Nester CM, Lambris JD, Smith RJ. Compstatin analog Cp40 inhibits complement dysregulation in vitro in C3 glomerulopathy. Immunobiology. 2015 Aug;220(8):993-8. doi: 10.1016/j.imbio.2015.04.001. Epub 2015 May 5. PMID 25982307
- [Background] Mastellos DC, Reis ES, Ricklin D, Smith RJ, Lambris JD. Complement C3-Targeted Therapy: Replacing Long-Held Assertions with Evidence-Based Discovery. Trends Immunol. 2017 Jun;38(6):383-394. doi: 10.1016/j.it.2017.03.003. Epub 2017 Apr 14. PMID 28416449
- [Derived] Hajishengallis G, Hasturk H, Lambris JD; Contributing authors. C3-targeted therapy in periodontal disease: moving closer to the clinic. Trends Immunol. 2021 Oct;42(10):856-864. doi: 10.1016/j.it.2021.08.001. Epub 2021 Sep 2. PMID 34483038